CLINICAL TRIAL: NCT01394588
Title: A Prospective Observational Trial of Continuous Glucose Monitoring Technology in the Perioperative Period During Cardiac Surgery
Brief Title: Continuous Glucose Monitoring Technology in the Perioperative Period During Cardiac Surgery
Status: Withdrawn | Type: Observational
Why Stopped: On further investigation, it was found that the continuous glucose monitors required a calibration period that precluded reliable data collection.
Sponsor: Yale University (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Robert Schonberger, Assistant Professor, Yale University
Other Study IDs: 1006006996
Record Dates: First submitted 2011-07-12; First posted 2011-07-14 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-05

CONDITIONS: Cardiac Surgery
Keywords: Cardiac Surgery; Perioperative Glucose Control

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiac Surgery Patients: Competent Adult Patients going for elective cardiac surgery.
  Interventions: Device: Use of continuous glucose monitor during surgery. ( Medtronic Minimed Guardian REALTime Continuous Glucose Monitor)

INTERVENTIONS:
Device: Use of continuous glucose monitor during surgery. ( Medtronic Minimed Guardian REALTime Continuous Glucose Monitor) — Use of continuous glucose monitor during surgery.
  Other Names: Medtronic Minimed Guardian REALTime Continuous Glucose Monitor

SUMMARY:
This is an observational study of continuous glucose monitoring technology during cardiac surgery. The investigators would like to develop data for descriptive analysis of a comparison of continuous glucose monitoring with a gold standard under the conditions of cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Competent adults scheduled for elective cardiac surgery.

Exclusion Criteria:

* Inability to consent, emergency surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Competent adults scheduled for elective cardiac surgery.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-08

CONTACTS AND LOCATIONS:
Overall Officials: Robert Schonberger, MD, Principal Investigator — Yale University